CLINICAL TRIAL: NCT01701271
Title: Evaluation of the Efficacy of the Cosmetic Lotion M.P.A.F. (Mixture of Paraffin, Alcohol and Fur) MEXIS PATENT in the Treatment of Androgenetic Alopecia by Decreasing of Hair Loss and Strengthening and Thickening of Hair in Males and Females.
Brief Title: Efficacy Study of a Cosmetic Lotion in the Treatment of Androgenetic Alopecia in Males and Females
Acronym: MEXISPATENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexis George (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEXIS-HAIR LOSS-STUDY 1.2012
Record Dates: First submitted 2012-10-01; First posted 2012-10-05 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Androgenetic Alopecia
Keywords: Baldness; Androgenetic Alopecia; Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volunteers (Experimental): 20 volunteers both men and women with an age between 18 and 70 years suffering from Androgenetic Allopecia in several types apply on the scalp drops of the hair loss prevention lotion
  Interventions: Other: Hair loss prevention lotion

INTERVENTIONS:
Other: Hair loss prevention lotion — For greatest problems 20 drops on the scalp per day for 3 months. For minor problems 10 drops on the scalp three times per week for 3 months.

SUMMARY:
The purpose of this study is to determine whether the Hair Loss Prevention Lotion named MEXIS, M.P.A.F., M6S PATENT is effective in the treatment of Androgenetic Alopecia.

DETAILED DESCRIPTION:
This study verifies whether the tested product has any efficacy in the treatment of Androgenetic Alopecia.

* The evaluated product (Hair Loss prevention Lotion) is called:MEXIS, MPAF, M6S PATENT.
* 20 volunteers both men and women suffering from hair loss both in parties and over the entire scalp with age between 18 and 70 years have been selected for this test .
* Samples of the product have been applied following their usual use: as they are.
* On the selecting volunteers have been used:

  1. The pull test by pulling with fingers of some hair and counting them to estimate the evolution of the pathology.
  2. A sebum-meter to check the presence of scales on the scalp.
  3. A polarized light video-camera to check the redness of the scalp and to have a picture of hair and scalp.
* Volunteers were also asked about:
* Fluffiness
* Sheen
* Itching
* Presence of scales on scalp
* Oily hair
* Product's acceptability
* The readings are taken at 0 time (basal value), after 15 days (t15), 30 days (t30), 45 days (t45), 45 days (t45), 60 days (t60) and 90 days (t90) by the experimenter in the medical studio. Then they analyzed and reported in a graph.
* Summarizing tables and graphs of the data were taken during experimentation.

ELIGIBILITY:
Inclusion Criteria:

* Good state of general health
* Suffering from hair loss
* No pharmacological treatment in progress
* Promise not to change the usual daily routine
* No atopy in the anamnesis

Exclusion Criteria:

* Illness
* Good state of hair
* Pharmacological treatment in progress
* Denial of the continuance of the usual daily routine
* Atopy in the anamnesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2001-02; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Marzatico, Monitor, Study Chair — Bio Basic EuropeResearch, Development and Dermo-Cosmetoligical Documentation
Locations (1):
- George Mexis, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on February 2001 at the University of studies of Pavia
Groups:
- Volunteers Evaluated: 20 volunteers both men and women with an age between 18 and 70 years suffering from Androgenetic Alopecia in several types apply on the scalp drops of the Hair Loss Prevention Lotion
Period: Overall Study
Arm/Group | Volunteers Evaluated
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Volunteers: 20 volunteers both men and women with an age between 18 and 70 years suffering from Androgenetic Alopecia in several types apply on the scalp drops of the Hair Loss Prevention Lotion
Arm/Group | Volunteers
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 44 (26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Italy | 20

OUTCOME MEASURES:

1. Primary Outcome: Change of the Amount of Hair Loss in a Pull Test
Description: Measurement of the decrease of hair loss by pull test and pulling some hair with the fingers.
  Measurements estimated and reported every 15 days. The Measure reports decrease in fallen hair
Time Frame: baseline and 90 days
Population: Good state of general health Suffering from hair loss No pharmacological treatment in progress Promise not to change the usual daily routine No atopy in the anamnesis
Measure: Mean (Full Range); unit: Fallen hair
Arm/Group | Volunteers
Number analyzed (Participants) | 20
Fallen hair | 2.75 [0.0 to 4.0]

2. Secondary Outcome: Change of Sebum on a Sebum-meter
Description: Measurements checked and reported every 15 days of the decrease of existing sebum on the scalp of the volunteers with a sebum-meter.
Time Frame: baseline and 90 days
Population: Good state of general health Suffering from hair loss
Measure: Mean (Full Range); unit: mg sebum/c^2
Arm/Group | Volunteers Evaluated
Number analyzed (Participants) | 20
mg sebum/c^2 | 8.8 [0 to 30]

3. Primary Outcome: Change of the Density of the Hair on a Polarized Light Video-camera as a Measure of Efficacy.
Description: Number of hair was assessed for each participant with a polarized light video-camera every 15 days for a total of 6 assessments
Time Frame: baseline and 90 days
Population: as for outcome 1
Measure: Mean (Full Range); unit: hairs/square inch
Arm/Group | Volunteers
Number analyzed (Participants) | 20
hairs/square inch | 2.75 [0.0 to 4.0]

ADVERSE EVENTS:
Description: No adverse events were assessed
Arm/Group | Volunteers
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No